CLINICAL TRIAL: NCT06172868
Title: Home Ventilatory Support in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R210861
Record Dates: First submitted 2022-08-08; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Sleep Apnea Syndromes in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study consist of children, who have used home ventilatory support during years 2010-2020 in Tampere University Hospital. The study will describe retrospectively different diagnoses and symptoms which will lead to home ventilatory support. We also study compliance to treatment and it's disanvantages. The prospective part of the study describes the quality of live of these children by using questionnaires (PedSQL).

ELIGIBILITY:
Inclusion Criteria:

- ICD-10 Code for Sleep apnea diagnose G47.3 AND G47.3 diagnose found from pediatric electronic patient records between years 2010-2020 OR Patient name found from pediatric multidisciplinary home respiratory team's clinical list

Exclusion Criteria:

* Age over 16
* Patient starting home ventilation after 31st December 2020 or treatment ending before 1st January 2010
* patients with sleep apnea but without home respiratory support treatment
* Only theophylline treatment
* High-flow oxygen therapy
* Age over 16 at treatment onset
* Never started treatment
* Treatment starting point and ending before year 2010

Max Age: 16 Years | Sex: All
Age Groups: Child
Study Population: 93 patients treated by a multidisciplinary paediatric home ventilatory support -team from January 2010 to December 2020 in Tampere University Hospital. The individuals were identified combining two sources: the team´s clinical list of patients and a database search from patient records with ICD-10 diagnose G47.3 (Sleep Apnea) in Pediatric Patient records.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient demographics of patients from 0 up to 16 years old treated by a multidisciplinary home respiratory support-team during January 2010 to December 2020 in Tampere University Hospital, Finland | 2022-2023
  Data included patient demographics
Number of patients with clinical characteristics | 2022-2023
  Data included underlying medical conditions and medications. The circumstances for home respiratory support onset, frequency of follow-up, complications, operative interventions to treat sleep apnea before and during period with home respiratory support were collected. The type of respiratory support (device, mode, interface) was recorded.

SECONDARY OUTCOMES:
The duration of treatment | 2022-2023
  The duration of treatment during January 2010 to December 2020 in Tampere University Hospital, Finland were collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Mervi Järvelä, Ilmajoki, Finland